CLINICAL TRIAL: NCT01010789
Title: Armodafinil in Binge Eating Disorder (BED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lindner Center of HOPE (Other)
Collaborators: Cephalon (Industry); University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cephalon_001
Record Dates: First submitted 2009-11-09; First posted 2009-11-10 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Binge Eating Disorder; Overweight; Obese
MeSH Terms: conditions — Binge-Eating Disorder; Overweight; Obesity | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Armodafinil (Experimental): Flexible dose 150-250mg/day
  Interventions: Drug: Armodafinil
- Mathing Placebo (Placebo Comparator)
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Armodafinil — flexible dose 150-250mg/day
  Arms: Armodafinil
Drug: Armodafinil — 150-250mg/day; flexible dose
  Arms: Armodafinil
Drug: Matching placebo — Placebo comparator
  Arms: Mathing Placebo

SUMMARY:
The purpose of this research study is to study the effectiveness, tolerability and safety of armodafinil in outpatients with binge eating disorder.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria: Criteria for entering this study will include all of the following:

1. Subjects will meet the DSM-IV-TR criteria for a diagnosis of binge eating disorder (BED) for at least the last 6 months. The DSM-IV-TR criteria are as follows:

   1. Recurrent episodes of binge eating. An episode of binge eating is characterized by both of the following: eating, in a discrete period of time (e.g., within any two hour period), an amount of food that is definitely larger than most people would eat in a similar period of time under similar conditions; and a sense of lack of control over eating during the episode (e.g., a feeling that one cannot stop eating or control what or how much one is eating).
   2. The binge eating episodes are associated with at least three of the following: eating much more rapidly than normal; eating until uncomfortably full; eating large amounts of food when not feeling physically hungry; eating alone because of being embarrassed by how much one is eating; feeling disgusted with oneself, depressed, or feeling very guilty after overeating.
   3. Marked distress regarding binge eating.
   4. The binge eating occurs, on average, at least two days a week for six months.
   5. The episodes of binge eating do not occur exclusively during the course of bulimia nervosa or anorexia nervosa.
2. In addition, subjects will report at least 3 binge eating days per week for the 2 weeks prior to randomization prospectively documented in take-home binge diaries. A binge eating day (or binge day) is a day during which at least one binge eating episode occurs.
3. Subjects will have a BMI ≥ 25. The subject population is expected to include overweight and obese individuals.
4. Men or women, through the ages of 18 and 65 years, inclusive.

Exclusion Criteria:

1. Have concurrent symptoms of bulimia nervosa or anorexia nervosa.
2. Women who are pregnant, lactating, or of childbearing potential who are not using adequate contraceptive measures. All female subjects who still have a uterus will have a negative pregnancy test prior to randomization.
3. Subjects who are displaying clinically significant suicidality or homicidality.
4. Subjects who have begun a new psychological (e.g., supportive psychotherapy, cognitive behavior therapy, interpersonal therapy) or weight loss (e.g., Weight Watchers, Overeaters Anonymous) intervention within the 3 months before study entry. Subjects who are receiving psychotherapy that was initiated prior to 3 months of the beginning of the study will be allowed to continue to receive their psychotherapy during the trial only if they agree to not make any changes to the frequency or nature of their psychotherapy during the course of the drug trial.
5. A DSM-IV-TR diagnosis of substance abuse or dependence (except nicotine abuse or dependence) within the 6 months prior to randomization.
6. A lifetime DSM-IV-TR history of psychosis, mania or hypomania, or dementia.
7. History of any psychiatric or personality disorder (eg, schizotypal and borderline) which might interfere with a diagnostic assessment, treatment, or compliance.
8. Clinically unstable medical disease, including cardiovascular, hepatic, renal, gastrointestinal, pulmonary, metabolic, endocrine or other systemic disease which could interfere with diagnosis, treatment, or assessment of BED. Subjects should be biochemically euthyroid to enter the study.
9. Have a history of any major cardiovascular event in the past 6 months, including unstable angina, acute myocardial infarction, coronary angioplasty, or stroke.
10. History of seizures, including clinically febrile seizures in childhood.
11. Have uncontrolled hypertension (>160/100) or tachycardia (heart rate >110).
12. Have an ECG with significant arrhythmias or conduction abnormalities, which in the opinion of the physician investigator preclude study participation.
13. Have clinically relevant abnormal laboratory results, specifically including hypokalemia.
14. Subjects who have a known allergy to armodafinil.
15. Subjects requiring treatment with any drug which might interact adversely with or obscure the action of the study medication. This includes warfarin, anticonvulsants, clonidine, theophylline, and pseudoephedrine.
16. Subjects who have received any psychotropic medications (other than hypnotics) within four weeks prior to randomization, including monoamine oxidase inhibitors, tricyclics, selective serotonin reuptake inhibitors, antipsychotics, mood stabilizers, or psychostimulants.
17. Subjects who have received investigational medications or depot neuroleptics within three months prior to randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-11; Primary Completion 2014-11 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is binge day frequency as assessed by take-home patient diary | 12 treatment weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Lindner Center of HOPE, Mason, Ohio, United States

REFERENCES:
- [Derived] McElroy SL, Guerdjikova AI, Mori N, Blom TJ, Williams S, Casuto LS, Keck PE Jr. Armodafinil in binge eating disorder: a randomized, placebo-controlled trial. Int Clin Psychopharmacol. 2015 Jul;30(4):209-15. doi: 10.1097/YIC.0000000000000079. PMID 26011779